CLINICAL TRIAL: NCT06507917
Title: Concordance and Acceptability of Self-screening Versus Screening by a Healthcare Professional for HPV, a Risk Factor for Anal Cancer, by Swab in People Living With HIV
Acronym: a-HPVVIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024/CHU/42; 2024-A01508-39 (Other: idRCB)
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: HPV Infection
Keywords: HPV; HIV; anal screening
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- self-swabbing first (Experimental): Group A self-swabbing then swabbing by a healthcare professional
  Interventions: Diagnostic Test: anal swabbing
- swabbing by a healthcare professional first (Active Comparator): swabbing by a healthcare professional and then self-swabbing
  Interventions: Diagnostic Test: anal swabbing

INTERVENTIONS:
Diagnostic Test: anal swabbing — anal swabbing

SUMMARY:
Anal canal cancers are on the increase in France, with around 2,000 new cases per year. These lesions can be detected by directed biopsies or smear tests.

The incidence rate of anal cancer is 30 times higher in people living with HIV than in the general population.

According to a recent study, the risk of anal cancer is highest in this population, but is also high in heterosexual men over 30 and women over 30. However, the proposal of a proctological examination in this population is not systematic.

In France, there is no HPV screening for people living with HIV, but there is a recommendation for proctology consultation in certain cases, notably for men who have sex with men (MSM) or for women with vaginal cervical lesions.

Several oncogenic HPV serotypes have been identified in the genesis of anal cancer. The serotype identified as the most carcinogenic is HPV-16 (89%).

This study will look at anal HPV screening in people over 30 living with HIV, thus including a population for which no screening is currently offered (heterosexual men living with HIV and women living with HIV without vaginal cervical lesions), and will assess the concordance and acceptability of self-screening versus screening by a healthcare professional as part of a comprehensive anal cancer screening strategy in this population.

ELIGIBILITY:
Inclusion Criteria:

Patient :

* living with HIV
* aged 30 or over
* resident on Reunion island and followed at the University Hospital of Reunion Island (the only follow-up center on the island)
* Able to perform anal self-sampling
* Able to answer a questionnaire
* Affiliated with or benefiting from a social security scheme
* Have given free, informed and signed consent

Exclusion Criteria:

* People with a previous anal swab less than 7 days old
* Persons with a known current diagnosis of anal cancer
* Persons deprived of liberty by judicial or administrative decision, minors, and persons under legal protection: guardianship or curators

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the concordance of HPV-16 genotype results between self-sampling and professional sampling. | 7 days
  HPV-16 genotype results for the sample

SECONDARY OUTCOMES:
Evaluate the concordance of results for other oncogenic HPV genotypes between self-sampling and professional sampling. | 7 days
  HPV oncogenic genotype results for the sample
To assess the preference of anal self-swabbing over anal swabbing performed by a healthcare professional. | 7 days
  visual scale from 0 (strongly disagree) to 10 (strongly agree)
Compare the overall satisfaction of the 2 anal samplings. | 7 days
  visual scale from 0 (poor) to 10 (very good).
Compare the proportion of adverse events (discomfort, pain, bleeding, itching) in the 2 groups. | 7 days
  discomfort, pain, bleeding, inconvenience after each swabbing
Compare the acceptability of anal self-swabbing versus anal swabbing performed by a healthcare professional. | 7 days
  composite score, constructed from the satisfaction scores, from which we subtract the average of the adverse event and shame scores, asked after each swab.
Evaluate the prevalence of anal HPV (including oncogenic HPV). | 7 days
  The proportion and prevalence of the various HPVs in the study population will be described.

CONTACTS AND LOCATIONS:
Locations (2):
- Reunion (2):
  - CHU de la Réunion Recherche Clinique, Saint-Denis
  - CHU de la Réunion Recherche Clinique, Saint-Pierre

IPD SHARING:
Plan to Share IPD: No